CLINICAL TRIAL: NCT04494542
Title: Sustained Low Efficiency Dialysis Versus Continuous Renal Replacement Therapy for Acute Kidney Injury in Critically Ill Cirrhotics-A Pilot Randomized Controlled Trial.
Brief Title: Sustained Low Efficiency Dialysis Versus Continuous Renal Replacement Therapy for Acute Kidney Injury in Critically Ill Cirrhotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-36
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Hybrid Renal Replacement Therapy; Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sustained Low Efficiency Dialysis (Experimental): Sustained Low Efficiency Dialysis
  Interventions: Procedure: Sustained Low Efficiency Dialysis (SLED)
- Continuous Renal Replacement Therapy (Active Comparator): continuous renal replacement therapy
  Interventions: Procedure: Continuous Renal Replacement Therapy

INTERVENTIONS:
Procedure: Sustained Low Efficiency Dialysis (SLED) — sustained low efficiency dialysis (SLED)
  Arms: Sustained Low Efficiency Dialysis
Procedure: Continuous Renal Replacement Therapy — Continuous Renal Replacement Therapy
  Arms: Continuous Renal Replacement Therapy

SUMMARY:
The current prospective pliot randomized controlled trial has been designed to demonstrate non-inferiority of sustained low efficiency dialysis (SLED) when compared to continuous renal replacement therapy in managing AKI in context of cirrhotics with septic shock who are hemodynamically unstable. The patients would be randomized 1:1 to either SLED or CRRT after screening for the inclusion and exclusion criteria.

DETAILED DESCRIPTION:
Aim & Objectives

Primary objective To study the efficacy of sustained low efficiency dialysis versus continuous renal replacement therapy in cirrhotics with septic shock and severe AKI

Secondary Objectives Effects on renal recovery rates in the two groups To assess the effects on 7-day and 28-day mortality Efficacy on Lactate Clearance Duration of mechanical ventilation and ICU stay Effect on systemic hemodynamics and reversal of shock Clearance of endotoxin and pro-inflammatory cytokines Effect on coagulation and endothelial function Improvement in SOFA scores at 48 hours and day 5

Methodology All included patients would be randomised to receive either continuous renal replacement therapy or sustained low efficiency dialysis (SLED) Patients with septic shock would be screened. Following this, patients meeting the inclusion and exclusion criteria will be screened and randomized to the two treatment groups. Standard criteria will be considered to define refractoriness to fluids and initiation of dialysis. Fluid management would be performed using the dynamic indices in patients on mechanical ventilation or using IVC diameter and passive-leg rasing in non-intubated patients. In all patients, baseline endotoxin activity assay and blood and urine sample will be stored for looking at the effect of therapy on cytokine profile (TNF alpha, IL-IB, IL6, IFN-gamma, MCP-1, IL-10 and ADAMTS and vWillebrand factor). Septic shock would be defined as a clinical construct of sepsis with persisting hypotension requiring vasopressors to maintain MAP>=65 mm of Hg and having a serum lactate >2 mmol/L despite adequate volume resuscitation. The blood flow rate, dialysis flow rate and need of ultrafiltration would be recorded for all enrolled patients. Subsequent sessions of therapy would be done as per requirement and recorded. The dose of vasopressor in norepinephrine equivalent would be recorded for all patients at enrolment as under

Study Population:

Patients with cirrhosis with septic shock and AKI requiring dialysis

Indications for initiation of dialysis

1. Metabolic acidosis with ph<7.2 or serum bicarbonate <15 mEq/lt
2. Hyperkalemia with serum potassium >5.5 Meq/L non-responsive to standard treatment
3. Oliguria with or without fluid overload (non-responsive to diuretics) with urine output of less than 0.5ml/kg/hr despite fluid resuscitation
4. Uremic complications (encephalopathy, pericarditis etc.)

Study Design:

* A randomized controlled study- Non-inferiority trial
* The study will be conducted on patients admitted to Department of Hepatology from June 2020 to December 2020 at ILBS, New Delhi
* Study group will comprise critically ill patients with cirrhosis with septic shock and AKI requiring dialysis

Study Period: The study will be conducted on patients admitted to Department of Hepatology from May 2020 to December 2020 at ILBS, New Delhi

Sample Size Calculation: The study will be designed as a pilot RCT with an aim to enrol 25 patients in each group. At completion a decision for termination versus continuation of the study would be taken.

Intervention: CRRT versus SLED until renal recovery

Renal recovery would be defined as increase in urine output to more than 400ml/day in patients with anuria, resolution of metabolic complications or spontaneous decline in urea and creatinine necessitating stopping dialytic support

Monitoring and Assessment: Hourly till the patient is in the intensive care then every 7 days until day 28

Statistical analysis

* All variables shall be expressed in mean (sd) or median (range)
* Variables will be compared by Mann- Whitney U test
* For Categorical variables we will use Chi-Square or Fisher's test
* Survival analysis will be done using Cox-proportional regression analysis

Actuarial probability of survival shall be calculated by Kaplan- Meier graph and compared by log- rank test.

Adverse Effects: Worsening of hypotension, bleeding any cardiac side-effects, worsening lactate, hypothermia, bradycardia

Stopping Rule: clinically relevant bleeding (i.e., transfusion requirements of at least 2 units of packed red cells), arrythmias (brady or tachyarryhthmias), poorly tolerated supraventricular arrhythmia related blood stream infections, development of electrolyte abnormalities hypokalemia, hypophosphatemia or hypomagnesemia refractory to medical management, renal recovery

ELIGIBILITY:
Inclusion Criteria:

- Critically ill cirrhotics with septic shock defined as need of vasopressors to maintain MAP> 65 mm Hg and lacate >2 mmol/L despite adequate fluid resuscitation with severe AKI meeting criteria for dialysis

Exclusion Criteria:

* Patients with age less than 18 years or more than 65 years
* Severe known cardiopulmonary disease (structural or valvular heart disease, coronary artery disease, COPD, CKD)
* Patients with ACLF
* Patients with cerebral edema
* Patients with refractory shock i.e. requiring norepinephrine or equivalent >0.5ug/kg/min
* Severe coagulopathy platelets <20,000 and INR >4
* Active Bleed (Mucosal or variceal)
* Pregnancy
* Patients with moderate-severe ARDS i.e. Pa02/Fio2 ratio <200
* Extremely moribund patients with an expected life expectancy of less than 24 hours
* Failure to give informed consent from family members.
* Patient enrolled in other clinical trials
* Patients with Hepatorenal Syndrome, post renal obstructive AKI, AKI suspected due to glomerulonephritis, interstitial nephritis or vasculitis based on clinical history and urine analysis
* Patients who have already been on hemodialysis before their arrival in the intensive care unit
* Patients with severe vasodilatation SVR <400 dyn·s/cm5 and/or lactate > 5 mmol/L

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Development of intradialytic hypotension i.e. decrease in defined as a decrease in systolic blood pressure by ≥20 mm Hg or a decrease in MAP by 10 mm Hg after initiation of dialysis | at 6 hours after dialysis initiation

SECONDARY OUTCOMES:
Mortality in both groups | Day 28
Duration of mechanical ventilation and ICU stay | Day 28
AKI recovery at day 14 | Day 14
Renal failure related death at day 7 | Day 7
Lactate clearance at 12 in both groups | 12 hours
Lactate clearance at 24 hours in both groups | 24 hours
Reversal of shock at 48 hours | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided